CLINICAL TRIAL: NCT06793605
Title: Community Burden of Mycoplasma Genitalium Infection and Its Implications for Test-and-treat Strategies
Brief Title: Community Burden of MG Infection
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ngai Sze WONG, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: MGMSM1
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Sexually Transmitted Infection (STI); Mycoplasma Genitalium Infection
Keywords: Mycoplasma genitalium; Chlamydia trachomatis; Neisseria gonorrhoeae; men who have sex with men
MeSH Terms: conditions — Sexually Transmitted Diseases; Homosexuality

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — urine specimen, rectal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective: To assess the burden and the transmission dynamics of Mycoplasma genitalium (MG) infection in men who have sex with men in Hong Kong.

Design and setting: involving a) a cross-sectional study (completion of an online self-administered survey, followed by self-sampling for testing in the laboratory, and performance of HIV self-test); b) a mathematical modelling study to simulate the transmission dynamics of MG infection and resistant MG infection and compare the impacts of test-and-treat strategies.

Participants: Around 920 men who have sex with men would be recruited

DETAILED DESCRIPTION:
Cross-sectional study: A total of 920 men who have sex with men aged 18 or above and normally living in Hong Kong would be recruited. Eligible participants would be asked to complete a self-administered online survey, submit self-collected urine specimen and rectal swabs for Chlamydia trachomatis, Neisseria gonorrhoeae, and Mycoplasma genitalium testing in the laboratory, and submit HIV self-test results.

Mathematical modelling study: A compartmental model would be constructed to simulate the transmission dynamics of MG infection and resistant MG infection, and analyse the impact of different test-and-treat strategies.

ELIGIBILITY:
Inclusion Criteria:

* men who have sex with men aged 18 or above, normally living in Hong Kong, and could communicate in written and spoken English or Chinese

Exclusion Criteria:

* cannot provide consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: men who have sex with men in Hong Kong
Sampling Method: Non-Probability Sample
Enrollment: 920 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
prevalence of MG infection | 1 year
  detection of MG infections in self-collected samples divided by the total number of samples collected
prevalence of MG resistance mutations | 1 year
  detection of MG resistance mutations macrolide/fluoroquinolone in MG positive samples divided by the total number of MG positive samples

SECONDARY OUTCOMES:
prevalence of CT infection | 1 year
  detection of CT infections in self-collected samples divided by the total number of samples collected
prevalence of NG infection | 1 year
  detection of NG infections in self-collected samples divided by the total number of samples collected
co-infection of STIs | 1 year
  number of co-infection of HIV, CT, NG, and/or MG
history of STI and HIV testing | ever
  number of self-reported history of STI and/or HIV testing at survey

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No